CLINICAL TRIAL: NCT01095198
Title: Randomized Controlled Trial of Vaginal Self Sampling for Human Papillomavirus to Increase Cervical Cancer Screening Participation
Brief Title: Randomized Trial of Vaginal Self Sampling for Human Papillomavirus (HPV)
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: McMaster University (Other)
Collaborators: Juravinski Cancer Centre Foundation (Other); Merck Frosst Canada Ltd. (Industry); Public Health Agency of Canada (PHAC) (Other Government)
Responsible Party: Alice Lytwyn, McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RCTself
Record Dates: First submitted 2010-03-29; First posted 2010-03-30 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-07

CONDITIONS: Human Papillomavirus Infection; Cervical Intraepithelial Neoplasia
Keywords: vaginal self collection; human papillomavirus (hpv); cervical intraepithelial neoplasia
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Dysplasia | interventions — Vaginal Smears

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2nd Reminder Letter (Active Comparator): 50% of study participants who are overdue for Pap testing and do not respond to initial reminder letter will be be mailed a standard second reminder letter
  Interventions: Other: 2nd reminder letter for Pap testing
- Offer of Vaginal Self Collection (Experimental): 50% of study participants who are overdue for Pap testing and do not respond to initial reminder letter will be selected to be mailed a second reminder letter and offer of vaginal self collection
  Interventions: Device: offer of vaginal self collection; Other: 2nd reminder letter for Pap testing

INTERVENTIONS:
Device: offer of vaginal self collection — Women assigned to the intervention group will be offered the opportunity to self collect a vaginal specimen for HPV testing. They will be sent a letter explaining that a study of self testing is being performed, and will invite her to participate in this study. The letter will state that, if the patient prefers, she can perform a vaginal self-test in addition to, or instead of Pap smear testing. Patients are told that they have the option of completing the self-test on their own or in their physician's office with the help of their physician or practice staff. The letter will be accompanied by a self collection kit consisting of: a swab and test tube, pamphlet (with written instructions and diagram outlining procedure), instructional DVD and return envelope.
  Other Names: flocked swab (Copan Diagnostics Inc.)
  Arms: Offer of Vaginal Self Collection
Other: 2nd reminder letter for Pap testing — Women in both groups will receive a letter informing them that they are due for cervical screening. This is a standard letter, and is signed by the patient's individual family physicians. It will advise the patient that this is the second reminder letter that she is due for cervical cancer screening, and will invite her to phone the physician's office to obtain an appointment for Pap testing.
  Other Names: reminder letter

SUMMARY:
Up to 30% of Canadian women do not participate in Pap smear screening for cervical cancer prevention despite many being members of family practices and having access to family physicians. One reason is reluctance to undergo pelvic examination.

The investigators purpose is to determine whether the offer of vaginal self sample collection for oncogenic human papillomavirus (HPV) testing increases participation in cervical cancer screening compared to repeat reminder for Pap smear testing among female family practice members who have not previously responded to invitations for Pap testing.

DETAILED DESCRIPTION:
Pap smear screening for cervical cancer precursors has substantially reduced the incidence of invasive cervical cancer in Canada. While regular Pap screening can give up to 90% protection against cervical cancer, about 30% of Canadian women do not participate in regular screening.

Pap screening in Ontario is opportunistic. There are women who have family doctors and regularly present for other medical issues at their physician's office but forego Pap smear testing.

Numerous studies have shown that women are able to self collect vaginal samples, and that these samples can be tested for the presence of oncogenic human papillomavirus. A recent meta-analysis showed that HPV testing through physician collected samples had a sensitivity of 80%-90% for detection of cervical intraepithelial neoplasia (CIN) 2 or worse, and a specificity of 86%-95%. In comparison, a meta-analysis of self collected vaginal samples tested for HPV showed a sensitivity of 74% and a specificity of 88%.

Studies have reported that women find self collection acceptable. However, we have found that many women are more comfortable if a health care professional is available to help if needed, and so this option should be provided for self-testing.

We are proposing a randomized controlled trial to see whether (a) the offer of a vaginal self collection kit together with a second reminder for Pap testing will increase cervical screening participation amongst "never-screened" and "hard to reach" women, as compared to (b) a second reminder letter alone.

ELIGIBILITY:
Inclusion Criteria:

* members of consenting family physicians identified through OSCAR EMR
* overdue for Pap smear testing
* have not presented for Pap smear screening after 1 reminder letter

Exclusion Criteria:

* currently attending colposcopy clinic
* institutionalized
* without a cervix

Ages: 35 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1440 (Estimated)
Dates: Start 2010-04; Primary Completion 2012-11 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
uptake of screening invitation | 18 months

SECONDARY OUTCOMES:
Cervical Intraepithelial Neoplasia (CIN) 3 identified | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Alice Lytwyn, MD, FRCPC, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada